CLINICAL TRIAL: NCT07342491
Title: A Multicenter Trial of the ACTG (Advancing Clinical Therapeutics Globally for HIV and Other Infections)
Brief Title: Trial of the ACTG (Advancing Clinical Therapeutics Globally for HIV and Other Infections)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A5413
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
Keywords: Antiretroviral Therapy (ART); Viral Persistence; HIV
MeSH Terms: conditions — HIV Infections | interventions — Dasatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: dasatinib (Experimental): 100 mg by mouth daily
  Interventions: Drug: Dasatinib
- Arm 2: Placebo (Placebo Comparator): Placebo for dasatinib
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dasatinib — will be administered as one 100 mg capsule (over-encapsulated tablet) orally once daily for 12 weeks
  Arms: Arm 1: dasatinib
Other: Placebo — Placebo for dasatinib will be administered as one placebo capsule (over-encapsulated tablet) orally once daily for 12 weeks
  Arms: Arm 2: Placebo

SUMMARY:
This study will test if the medicine dasatinib can lower the hidden amount of HIV in the body, called the HIV "reservoir." It will also check if dasatinib is safe and easy to take for people living with HIV who have a suppressed viral load while on antiretroviral therapy (ART). Adults 18 years or older who have been on ART for at least 48 months and have had a suppressed HIV-1 viral load for at least 36 months may be able to join.

People will be randomly assigned to take dasatinib 100 mg by mouth once a day or a look-alike substance with no drug, called a placebo, for 12 weeks. Neither participants nor researchers will know who gets which (double-blind). The study team will do regular health checks and blood tests to track safety, tolerability, the HIV reservoir, and changes in immune cells.

The study lasts 36 weeks total: 12 weeks of treatment and 24 weeks of follow-up, with clinic visits and possible phone calls. Fourteen people will take part; eight will get dasatinib and six will get placebo. Dasatinib may lower the HIV reservoir, but this is not guaranteed. All medicines can cause side effects, called adverse events (AE). The study team will watch closely and provide medical support. Joining is your choice, and you can leave at any time. If you leave, the team will talk with you about next steps for your care.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Active antiretroviral therapy received continuously for 48 months (or longer)
* CD4+ cell count >450 cells/mm3 obtained within 12 months prior to study entry
* Plasma HIV-1 RNA level below the lower limit of quantification within 90 days prior to study entry
* Plasma HIV-1 RNA levels below the lower limit of quantification for >36 months at time of study entry
* The following laboratory values obtained within 90 days prior to entry:

  * Absolute neutrophil count (ANC) above the lower limit of normal
  * Hemoglobin above the lower limit of normal
  * Platelet count above the lower limit of normal
  * Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), and alkaline phosphatase <1.5 x ULN
  * Total bilirubin <1.5 x ULN
  * Negative hepatitis B virus (HBV) surface antigen (HBsAg)
  * Negative HBV core antibody with one exception: individuals with positive HBV core antibody and HBV surface antibody are eligible for enrollment
  * Negative hepatitis C virus (HCV) antibody (anti-HCV) or, if the anti-HCV is positive, a negative HCV RNA PCR
  * Estimated glomerular filtration rate (eGFR) >70 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) 2021 equation or serum creatinine <1.2 x ULN
* QTc interval <450 milliseconds on EKG performed at screening visit
* Women who are able to become pregnant must have a negative serum or urine pregnancy test at screening and within 48 hours prior to study entry
* Individuals (male or female) who are having sex that could lead to pregnancy, must agree to use at least two effective means of contraception when engaging in sexual activities that can result in pregnancy, from the time of enrollment through 60 days following the last dose of dasatinib
* Able to swallow pills without difficulty.
* Ability and willingness of participant or legally authorized representative to provide informed consent
* Ability and willingness of participant to continue same ART regimen throughout the study

Exclusion Criteria:

* Pre-ART viral load known to be <2000 copies/mL (HIV controller)
* Known to have initiated ART during acute HIV infection
* Presence of a drug-resistant virus with no alternative ART regimens available in the event that current ART regimen becomes compromised as a result of this study
* Current pregnancy or breastfeeding or pregnancy planning during study participation
* Recent hospitalization or surgery within 90 days prior to entry
* Recent infection requiring intravenous antibiotics within 90 days prior to entry
* Any evidence of hepatic impairment
* Any known prior (lasting >180 days) or current history of gastrointestinal-related diseases
* Active malignancy including myelodysplastic syndrome or myeloproliferative disease.
* Any known prior (lasting >180 days) or current history of hematologic illness
* Any known prior (lasting >180 days) or current history of cardiac-related diseases
* Untreated hypothyroidism
* Treatment for TB within the past 90 days.
* Current respiratory disease requiring supplemental oxygen
* Exposure to any systemic immunomodulatory drug (including maraviroc) in the 16 weeks prior to study entry
* Exposure to anticoagulant or anti-platelet medications in the 16 weeks prior to study entry
* Active use of medications known to prolong the QT interval
* Known family history of Long QT Syndrome in a first-degree relative (i.e., parent, offspring, or sibling)
* Active use of medications known to moderately or strongly induce or inhibit CYP3A4, including ART regimens that contain protease inhibitors, efavirenz, etravirine, or cobicistat at the time of screening or study entry
* Current substance use which is likely to interfere with the conduct of the study
* Anticipated conflict or inability to attend and complete all protocol-scheduled study visits and assessments
* Known allergy/sensitivity or any hypersensitivity to components of dasatinib or its formulation
* Active use of azithromycin, Ondansetron, Pentamidine at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-11-25 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Change in intact HIV-1 reservoir size | Baseline and week 12
  Change in the intact HIV-1 reservoir from baseline to week 12, measured by the Intact Proviral DNA Assay (IPDA), or the best available assay at the time of testing if IPDA is not available.
Number of Study treatment-related adverse events | From first dose through week 36
  Occurrence of any study treatment-related serious adverse event (SAE), any Grade 2 or higher adverse event (AE), or any AE that leads to permanent discontinuation of study treatment, regardless of grade.

SECONDARY OUTCOMES:
Anti-proliferative effects after 1 week of dasatinib | Baseline and week 1
  Change in immune cell proliferation after 1 week of dasatinib, compared with baseline. Proliferation will be assessed in CD4+ and/or CD8+ T cells using standard markers or assays
Changes in T cell subset composition and cellular Ki-67 expression | Baseline to week 12
  Changes from baseline to week 12 in T cell subset composition and Ki-67 expression.
Changes in HIV-1 cell-associated RNA transcripts in total CD4+ T cells | Baseline to week 12
  Measured in total CD4+ T cells
Changes in low-level plasma viremia (single-copy assay) | Baseline to week 12
  Measured using the single-copy assay

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwestern University CRS (Site # 2701), Chicago, Illinois
  - 2501, Case CRS, Cleveland, Ohio
  - 1401, University of Washington Positive Research CRS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the ACTG (Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections) by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG (Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections).
  * For what types of analyses? To achieve aims in the proposal approved by the ACTG.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.